CLINICAL TRIAL: NCT06709326
Title: APACA-Apheresis/acoustophoresis and Molecular Characterization of Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: APACA
Record Dates: First submitted 2023-03-17; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Androgen Antagonists

STUDY DESIGN:
Intervention Model Description: Three groups of research subjects
  1. Primary metastatic prostate cancer
  2. PSA relapse
  3. Healthy research subjects
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Primary metastatic prostate cancer (Experimental): Men who have not previously received treatment for prostate cancer.
  Interventions: Diagnostic Test: Apheresis; Other: Androgen deprivation therapy
- PSA relapse (Experimental): Men with PSA recurrance after surgery.
  Interventions: Diagnostic Test: Apheresis; Diagnostic Test: Anti androgen therapy
- Healthy research subjects (Other): Control group to distinguish tumor-specific changes from normal signals.
  Interventions: Diagnostic Test: Apheresis

INTERVENTIONS:
Diagnostic Test: Apheresis — Isolate tumor cells, immune cells, exosomes and cell free DNA from the blood by a clinically used method of whole blood volume filtration, apheresis, and subsequent separation of blood components using novel techniques, such as acoustophoresis and other experimental protocols.
Other: Androgen deprivation therapy — Apheresis will be performed before initiation of systemic therapy (androgen deprivation therapy) and 4 weeks after. Androgen deprivation therapy is treatment as per clinical routine and not part of the protocol.
  Arms: Primary metastatic prostate cancer
Diagnostic Test: Anti androgen therapy — Apheresis will be performed before initiation of systemic therapy (anti androgen therapy). Anti androgen therapy is treatment as per clinical routine and not part of the protocol.
  Arms: PSA relapse

SUMMARY:
The goal of this clinical study is to to improve diagnosis, follow-up and treatment for patients with disseminated prostate cancer.

The aim is to isolate tumour cells before image diagnostic methods find the metastases. In addition, investigators will use this method to characterise the tumour cells at the "single-cell" level to understand both the metastasis process, early resistance mechanisms and thus find new treatment targets to optimise individualised treatment.

Research subjects who either have disseminated disease at diagnosis or have recurrence after surgery (with minimal dissemination) will be included. A control population of young men without cancer will also be recruited to distinguish tumor-specific changes from normal signals using these new methods.

DETAILED DESCRIPTION:
In this prospective clinical study, led by Umeå University, all research subjects will undergo apheresis and subjects with cancer will also undergo multiple radiological examinations to both identify apheresis and subsequent experimental protocols for isolation of tumor cells, immune cells and other components from the blood. The goal is to increase the sensitivity of identifying circulating tumor cells in early-stage metastatic prostate cancer for molecular characterization without biopsies of metastases. By doing this on multiple occasions in primary metastatic prostate cancer, investigators will identify early resistance mechanisms to given treatment and also investigate immune changes to standard treatment of metastatic prostate cancer (castration). Through qualitative approach, investigators will identify healthy and risk factors for managing the diagnosis of metastatic prostate cancer and the experience of undergoing apheresis to identify circulating tumor cells (CTC) in the blood, with the aim of identifying possible risks for mental health with this research.

ELIGIBILITY:
Inclusion Criteria:

-The patient (arm 1 and arm 2) must have a health status that minimises the already low risks of the apheresis treatment, have the logistical possibilities to come to the visits according to the study and be planned for treatment according to standard treatment in Sweden today.

For arm 1, 2 and 3:

* Venous blood vessels enabling apheresis
* ECOG-performance status 0-2
* Concentration of av potassium, calcium and magnesium in blood within normal range
* Testosterone>1,7 nmol/L
* Hb>90 g/L
* TPK >50x10exp9 /L
* LPK >1x10exp9 /L
* Bilirubin <1,4 x upper limit for normal (unless the subject suffers from Gilberts disease)
* ALAT or ASAT <2,4 x above limit for normal
* Creatinine <2 mg/dL (<177µmol/L)

Additional inclusion criteria for Arm 1 - Metastatic prostate cancer

One of the following criteria:

* PSA >100ng/ml
* Skeletal metastases with high risk of prostate cancer (regardless of PSA-value)

Additional inclusion criteria for Arm 2 - PSA relapse after operation

All of the three following criteria must be fulfilled:

* Prostatectomy
* PSA >0.2ng/ml
* PSA doubling time <18 months (according to www.mskcc.org/nomograms/prostate/psa_doubling_time)

Additional inclusion criteria for Arm 3 - Healthy research subjects (control group)

All of the following two criteria must be fulfilled:

* Previously healthy (no ongoing medication)
* No history of cancer

Exclusion Criteria for arm 1, 2 and 3:

* Overall, research subjects must not have any other cancer disease or risk factors for undergoing apheresis treatment
* Weight <50 kg
* Medical castration last 6 months (or previous surgical castration)
* Antiandrogen treatment in the last 6 months
* Previous myocardial infarction, stroke, chronic heart failure, atrial fibrillation or multiple deep vein thromboses
* Heart rate <45
* Systolic blood pressure below 100
* Ongoing diagnosed chronic inflammation

Ages: 18 Years to 81 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2020-09-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Identify circulating tumor cells (CTC) for molecular characterization | At inclusion in the study and after 4 weeks of treatment.
  Identification of circulating tumor cells will be accomplished by RNA-based phenotyping using lineage specific transcripts.
Differentiated gene expression in CTCs before and after treatment start | At inclusion in the study and after 4 weeks of treatment.
  To find resistance mechanisms by deep molecular characterization of CTC before and after treatment start to identify up and down regulations of genes in paired samples.
Phenotypical changes of immune cells due to anti-androgen treatment | At inclusion in the study, after 4 weeks of treatment, after 3, 6 and 12 months of treatment.
  Broad molecular characterization of immune cells before initiation of treatment and at different time points after anti-androgen treatment

SECONDARY OUTCOMES:
Progression free survival | Within 24, 48 and 72 months respectively
  Time to progression defined as PSA relapse or new metastasis or prostate cancer death, which ever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Josefsson, MD, PhD, Principal Investigator — Department of surgical and perioperative sciences, Urology, Umeå University
Locations (1):
- Department of surgical and perioperative sciences, Umeå university, Umeå, Norrlands University Hospital, Sweden